CLINICAL TRIAL: NCT06757998
Title: On-lay Versus Pre-peritoneal Hernioplasty in Incisional Lumbar Hernia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali fathy Ali, AFAli, Assiut University
Other Study IDs: Hernioplasty in lumbar hernia
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Lumbar Hernia
MeSH Terms: conditions — Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mesh — Compare between On-lay versus pre-peritoneal hernioplasty in incisional lumbar herni

SUMMARY:
To compare between the outcome of on-lay and pre-peritoneal techniques of hernioplasty in incisional lumbar hernia repair.

DETAILED DESCRIPTION:
Lumbar hernia is found as a challenge even in the era of advanced medicine, due to its rarity which complicate its diagnosis and treatment[1]. Lumbar hernia is the protrusion of an organ intra-peritoneal or extra-peritoneal tissue through a congenital or acquired defect in the posterolateral abdominal wall[2]. Incisional Lumbar hernia is among the types of lumbar hernia that accounts for 25% of cases[3]. Post abdominal surgeries, the tissue strength can only regain 80% of its maximum tensile power under perfect conditions. Thus, each abdominal surgery is a predisposing factor for lumbar incisional hernia [4] Primary closure of the defect with sutures, has proven to have a high failure rate so the integration of the mesh in hernia repair has significantly flattened the recurrence curve. Taking the advantage of Laplace's law, the mesh aims to reinforce or bridge the defect and distribute the intra-abdominal pressure across the entire synthetic sheet rather than just the defect. [5] The two most used mesh placing techniques are on-lay and pre-peritoneal. Each method has its benefits and drawbacks. [6] Some surgeons outweigh the on-lay technique to avoid extensive dissection. Thus, it is a faster and easier technique; nevertheless, there are several local wound issues. [7] The pre-peritoneal method allows the surgeon to apply the mesh posterior to the fascial plane in front of the peritoneum. The latter technique is gaining popularity with time [8]

Literature are deficient in comparing on-lay and pre-peritoneal technique in the repair of incisional lumbar hernia.

ELIGIBILITY:
Inclusion Criteria:

* Incisional lumbar hernia
* Recurrent lumbar hernia
* Age more than 16 years old

Exclusion Criteria:

* Complicated lumbar hernia (irreducible, obstructed, strangulated hernia)
* Denovo lumbar hernia

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: • Conventional Sample size of about 30 Cases about 15 cases of each group
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-29 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Short term complications (Recurrence, Postoperative Seroma and skin infection.) | Two months